CLINICAL TRIAL: NCT00460590
Title: A Phase I Study Evaluating the Safety and Immunogenicity of a New TB Vaccine MVA85A, in Healthy Volunteers With no Evidence of Infection With Mycobacterium Tuberculosis, in Cape Town
Brief Title: Safety and Immunogenicity of MVA85A, in Healthy Volunteers in Cape Town
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: University of Cape Town (Other)
Responsible Party: Dr Helen McShane, University of Oxford
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TB008
Record Dates: First submitted 2007-04-13; First posted 2007-04-16 (Estimated); Last update posted 2008-08-07 (Estimated); Status verified 2008-06

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; TB; MVA 85A
MeSH Terms: conditions — Tuberculosis | interventions — MVA 85A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): 12 adults with prior BCG
  Interventions: Biological: MVA 85A
- 2 (Experimental): 12 adults without prior BCG
  Interventions: Biological: MVA 85A
- 3 (Experimental): 12 Adolescents
  Interventions: Biological: MVA 85A

INTERVENTIONS:
Biological: MVA 85A — ID vaccine

SUMMARY:
This study is designed to evaluate the safety of MVA85A in healthy volunteers in Cape Town. We have shown that MVA85A is safe and immunogenic in both a mycobacterially naïve population in the UK and in a more mycobacterially exposed population in The Gambia. The studies described here will be to assess the safety of MVA85A in 2 groups of adults, those with and without prior BCG vaccination. Once safety data has been obtained in these 2 groups, we will assess the safety of MVA85A in adolescents who have been previously vaccinated with BCG.

DETAILED DESCRIPTION:
This is an open label Phase I safety study of a single intradermal injection of 5 x 107pfu MVA85A, when administered to healthy subjects with no evidence of infection with M.tb

Sample size:

This is an observational and descriptive safety study, 12 subjects with evidence of prior BCG vaccination and 12 adults with no evidence of prior BCG vaccination will be recruited and vaccinated with MVA85A. This sample size should allow determination of the magnitude of the outcome measures, especially of serious and severe adverse events rather than aiming to obtain statistical significance. Once three month follow-up of these two arms of the study is complete, we will recruit 12 adolescent school children (aged 12-14) and assess the safety and immunogenicity of a single immunisation with MVA85A in this group.

Rules for progression from adult studies to adolescents:

1. No increased incidence in local and systemic side-effects compared with trials with MVA85A in Oxford and The Gambia.

   In the trials in the UK and The Gambia, all volunteers experience some mild local side-effects for 1-4 days after vaccination.

   Approximately two- thirds of volunteers experience some mild systemic side-effects in the first 24 hours after vaccination. These are self-limiting and all spontaneously resolve.

   These side-effects are consistent with data from use with other recombinant MVAs expressing other antigens (Moorthy VS et al, 2003).
2. Immune responses measured 1 week after vaccination. We see strong immune responses 1 week after vaccination in the Oxford and Gambian volunteers (McShane et al, 2004). We do not know how long the responses in the South African volunteers will last for, but we would expect to see the induction of significant (compared with baseline) immune responses as measured by the ex-vivo Elispot assay, 1 week after vaccination

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 50 years (for the first 2 arms)
* Healthy adolescents (aged 12-14) for the third arm of the study
* Screening Elispot negative (less than 17 spots/million PBMC) in all 3 ESAT6 pools and all 3 CFP10 pools
* Mantoux test <15mm (<10mm if BCG naïve)
* CXR normal with no evidence of active or past TB
* For females only, willingness to practice continuous effective contraception during the study and a negative pregnancy test on the day of vaccination
* Agreement to refrain from blood donation during the course of the study
* Written informed consent
* Willingness to undergo an HIV test

Exclusion Criteria:

* Any deviation from the normal range in biochemistry or haematology blood tests or in urine analysis as defined in Appendix I
* Mantoux >15mm
* Prior receipt of a recombinant MVA or Fowlpox vaccine
* Use of any investigational or non-registered drug, live vaccine or medical device other than the study vaccine within 30 days preceding dosing of study vaccine, or planned use during the study period
* Administration of chronic (defined as more than 14 days) immunosuppressive drugs or other immune modifying drugs within six months of vaccination. (For corticosteroids, this will mean prednisolone, or equivalent, 0.5 mg/kg/day. Inhaled and topical steroids are allowed.)
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection and asplenia
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g. egg products
* Evidence of cardiovascular disease
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of diabetes mellitus
* Chronic or active neurological disease requiring ongoing specialist or medical supervision
* Chronic gastrointestinal disease requiring ongoing specialist or medical supervision
* History of > 2 hospitalisations for invasive bacterial infections (pneumonia, meningitis)
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
* Seropositive for hepatitis B surface antigen (HBsAg)
* Seropositive for hepatitis C virus (antibodies to HCV)
* Evidence of serious psychiatric condition
* Any other on-going chronic illness requiring hospital specialist or medical supervision
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Pregnant or lactating female
* Female who is willing or intends to become pregnant during the study
* Any history of anaphylaxis in reaction to vaccination
* Inability to give informed consent
* PI assessment of lack of willingness to participate and comply with all requirements of the protocol
* Any other finding which in the opinion of the investigator would significantly increase the risk of having an adverse outcome from participating in this protocol

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2005-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
To assess the safety of a single intradermal injection of 5 x 107pfu MVA85A, when administered to healthy subjects. The specific endpoints for safety and reactogenicity will be actively and passively collected data on adverse events (AEs). | year

SECONDARY OUTCOMES:
To assess the immunogenicity of a single vaccination with MVA85A in healthy subjects. The specific endpoints for immunogenicity will be markers of cell-mediated immunity as outlined above | year

CONTACTS AND LOCATIONS:
Overall Officials: Greg Hussey, Professor, Principal Investigator — University Cape Town
Locations (1):
- University Cape Town, Cape Town, South Africa

REFERENCES:
- [Derived] Tanner R, Kakalacheva K, Miller E, Pathan AA, Chalk R, Sander CR, Scriba T, Tameris M, Hawkridge T, Mahomed H, Hussey G, Hanekom W, Checkley A, McShane H, Fletcher HA. Serum indoleamine 2,3-dioxygenase activity is associated with reduced immunogenicity following vaccination with MVA85A. BMC Infect Dis. 2014 Dec 3;14:660. doi: 10.1186/s12879-014-0660-7. PMID 25466778
- [Derived] Hawkridge T, Scriba TJ, Gelderbloem S, Smit E, Tameris M, Moyo S, Lang T, Veldsman A, Hatherill M, Merwe Lv, Fletcher HA, Mahomed H, Hill AV, Hanekom WA, Hussey GD, McShane H. Safety and immunogenicity of a new tuberculosis vaccine, MVA85A, in healthy adults in South Africa. J Infect Dis. 2008 Aug 15;198(4):544-52. doi: 10.1086/590185. PMID 18582195